CLINICAL TRIAL: NCT06242041
Title: The Effect of Potassium Lowering Drugs on Cardiac Electrical Stability in Hemodialysis
Brief Title: The Effect of Potassium Lowering Drugs on Cardiac Electrical Stability in Hemodialysis Patients (ART Study)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Li LIU, Medical Doctor, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2022CR08
Record Dates: First submitted 2024-01-28; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-01

CONDITIONS: Potassium Imbalance; Cardiac Arrhythmia; Dialysis; Complications
Keywords: Hyperkalemia; Chronic kidney disease; Maintenance hemodialysis; cardiac electrical stability; New oral potassium-lowering drugs; T wave alternans
MeSH Terms: conditions — Arrhythmias, Cardiac; Hyperkalemia; Renal Insufficiency, Chronic | interventions — Renal Dialysis

STUDY DESIGN:
Intervention Model Description: Treatment group: routine treatment, and oral potassium reduction by SZC on non-dialysis day.
  Control group: routine treatment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Routine treatment, and on the non-dialysis day, sodium zirconate silicate is given four times a week, starting from 5g/ day each time, and the blood potassium before dialysis is maintained at 4.0-5.0mmol/L, which can be adjusted by 10g/ week each time, and the highest dose can be increased to 80g/ week.
  Interventions: Drug: sodium zirconium cyclic silicate
- Control group (Placebo Comparator): Routine treatment.
  Interventions: Drug: sodium zirconium cyclic silicate

INTERVENTIONS:
Drug: sodium zirconium cyclic silicate — On the non-dialysis day, the drug was given to patients in the treatment group, four times a week, starting from 5g/day each time, and the blood potassium before dialysis was maintained at 4.0-5.0mmol/L, which could be adjusted at 10g/week each time, and the highest dose could be increased to 80g/ week.
  Other Names: hemodialysis

SUMMARY:
This study is a multicenter, prospective and randomized controlled study. The experiment includes a 1-week screening period (1 week before dialysis) and a 7-week treatment period (1-4 weeks of dose drip period and 5-7 weeks of evaluation period). During the screening period, all patients were randomly divided into the control group and the treatment group. On the non-dialysis day of the treatment period, the treatment group was given a certain dose of sodium zirconium silicate, and the blood potassium value was measured before and after each dialysis to maintain the blood potassium at 4.0-5.0mmol/L before dialysis. At the same time, 12-lead ECG and 24-hour Holter were completed at the first and last dialysis during the treatment period, and finally the ECG stability and its relationship with blood potassium were evaluated.

DETAILED DESCRIPTION:
1. Screening period (1 week before administration):

   After 72 hours without dialysis treatment and before dialysis for the first time, complete the set 1 of laboratory inspection group, including hemoglobin, white blood cells, platelets, serum creatinine, urea nitrogen, alanine aminotransferase, aspartate aminotransferase, albumin, potassium, calcium, magnesium and bicarbonate. After dialysis, complete the set 2 of laboratory inspection group, including urea nitrogen and potassium. According to the ratio of 1: 1, the patients were randomly divided into control group (routine treatment) and experimental group (sodium zirconium silicate was given on the basis of routine treatment).
2. Dose drops period (1st week to 4th week):

Blood samples are collected before and after dialysis for the first time every week to complete the set 3 of laboratory inspection group, including: potassium, and the dosage of SZC is adjusted according to the blood potassium value, which is administered on non-dialysis days, four times a week, starting from 5g/day each time, and the blood potassium before dialysis is maintained at 4.0-5.0mmol/L, which can be adjusted at 10g/week each time, and the highest dosage can be increased to 80g/week.

1. If the blood potassium is higher than 5.0mmol/L during the follow-up, the amount of SZC can be gradually increased to 30-80g per week.
2. If during the follow-up, the blood potassium before dialysis is lower than 5mmol/L, and the potassium concentration of dialysate is raised to 3mmol/L, other ion concentrations remain unchanged, including calcium, bicarbonate, sodium and magnesium. If the blood potassium is still below 5mmol/L in the follow-up, the SZC will be reduced to 10g per week. If the blood potassium is lower than 4.0mmol/L in the follow-up, stop the experiment.

In the first week of drip period, 12-lead ECG and Holter were completed on the day of dialysis.

3.Evaluation period (week 5 to week 7): At the end of the experiment, blood was collected before the last dialysis to complete the laboratory inspection group set 1, and the 12-lead electrocardiogram was improved and Holter was worn, while blood was collected after dialysis to complete the laboratory inspection group set 2.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years old.
2. ESKD received hemodialysis treatment three times a week for more than 3 months.
3. After a long interval, before dialysis, the serum potassium was≥5.0mmol/L and was examined for two months in a row.
4. Screening patients with serum potassium≥5.0mmol/L before dialysis.

Exclusion Criteria:

1. poor compliance with dialysis treatment.
2. Acute myocardial infarction, acute coronary syndrome, stroke, epilepsy or thromboembolism (such as deep vein thrombosis or pulmonary embolism, but excluding hemodialysis pathway thrombosis) occurred within 12 weeks before the screening date.
3. Hypokalemia (blood potassium<3.5mmol/L), hypocalcemia (blood calcium<2.1mmol/L), hypocalcemia (blood magnesium<0.7mmol/L) or severe acidosis (blood bicarbonate<16mmol/L) occurred within 4 weeks before the screening date.
4. Severe hematological abnormalities: white blood cells>20×10^9/L, platelets≥450×10^9/L.
5. Rhabdomyolysis was diagnosed 4 weeks before screening.
6. Taking lactulose, rifaximin or other unabsorbed antibiotics to treat hyperammonemia within 7 days before taking the first medicine.
7. Patients cannot take sodium zirconium silicate orally.
8. The patient is allergic to sodium zirconium silicate or other components of the drug.
9. The life expectancy of patients is less than 1 year.
10. Patients during pregnancy and lactation.
11. Female patients preparing for pregnancy during the study period.
12. Participated in clinical research of other drugs in the month before screening.
13. Persons who have lost their autonomous capacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Estimated)
Dates: Start 2022-02-14 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Potassium lowering effect | 7 weeks.
  The decrease of serum potassium in the treatment group before dialysis after using sodium zirconium silicate was compared with that in the control group.
Changes of ECG stability during dialysis. | 7 weeks.
  To compare the changes of ECG activity between the treatment group and the control group during dialysis after potassium reduction treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University first hospital hemodialysis center, Beijing, Beijing Municipality, China